CLINICAL TRIAL: NCT02903498
Title: Phase II Study of the Maintenance Treatment of UFT (Uracil and Tegafur) After First-line
Brief Title: The Maintenance Treatment of UFT in Advanced Gastric Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, Xiaodong Zhu, MD, PhD, Fudan University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: UFT maintenance in GC
Record Dates: First submitted 2016-09-04; First posted 2016-09-16 (Estimated); Last update posted 2016-10-12 (Estimated); Status verified 2016-10

CONDITIONS: Gastric Cancer
Keywords: disease control survival
MeSH Terms: conditions — Stomach Neoplasms | interventions — Tegafur

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- UFT treatment (Experimental): Uracil and Tegafur
  Interventions: Drug: UFT
- comparator (No Intervention): no treatment, follow-up at regular time

INTERVENTIONS:
Drug: UFT — UFT 360mg/m2 qd po d1-14, q3w
  Other Names: Uracil and Tegafur
  Arms: UFT treatment

SUMMARY:
The purpose of this study is to evaluate the efficacy and tolerability of the maintenance treatment of tegafur-uracil (UFT) after the standard first-line chemotherapy in advanced gastric cancer.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed advanced or metastatic adenocarcinoma of the stomach
* ECOG PS 0-2
* At least one measurable or evaluable lesion in the first-line chemotherapy (5-FU based regimen: ECF/EOF/EOX/FOLFOX/XELOX) with the efficacy evaluation of non-PD
* Adequate hepatic,renal,heart, and hematologic functions (platelets ≥75×109/L, neutrophil≥1.5×109/L, hemoglobin≥80 g/L, serum creatinine ≤1.5mg/dl, total bilirubin ≤1.5mg/dl, and serum transaminase≤2.5×the ULN)

Exclusion Criteria:

* Receiving more or more than 2 regimens of chemotherapy
* Pregnant or lactating women
* Concurrent cancer
* History of other malignancies except cured basal cell carcinoma of skin and carcinoma in-situ of uterine cervix
* Neuropathy, brain, or leptomeningeal involvement
* Clinically relevant coronary artery disease or a history of a myocardial infarction within the last 12 months or high risk/uncontrolled arrhythmia
* Uncontrolled significant comorbid conditions and previous radiotherapy

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 58 (Actual)
Dates: Start 2009-08; Primary Completion 2016-06 (Actual); Study Completion 2016-09 (Actual)

PRIMARY OUTCOMES:
Progression Free Survival (PFS) | six weeks
  PFS is calculated from the start of treatment to disease progression or death

SECONDARY OUTCOMES:
Overall Survival (OS) | six weeks
  OS is calculated from the start to treatment to the death
Number of Participants with Adverse Events | six weeks

CONTACTS AND LOCATIONS:
Overall Officials: Xiaodong Zhu, Principal Investigator — Fudan University